CLINICAL TRIAL: NCT03751540
Title: Ultrasound-guided Oblique Subcostal Transversus Abdominis Plane Block Versus Serratus Intercostal Plane Block Plus Rectus Sheath Block; in Laparoscopic Cholecystectomy
Brief Title: Retrospective Evaluation of Plane Blocks in Laparoscopic Cholecystectomy
Status: Completed | Type: Observational
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Asst. Prof. Serkan Tulgar, M.D., associated professor, Maltepe University
Other Study IDs: Blocks in LC
Record Dates: First submitted 2018-11-19; First posted 2018-11-23 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OSTAP: Data of patients (performed oblique subcostal transversus abdominis plane-OSTAP- block for postoperative analgesia in laparoscopic cholecystectomy) will be collected.
  Interventions: Procedure: ostap
- SIPB plus rectus sheath block: Data of patients (performed serratus intercostal plane block-SIPB- plus rectus sheath block for postoperative analgesia in laparoscopic cholecystectomy) will be collected.
  Interventions: Procedure: SIPB plus rectus sheath block

INTERVENTIONS:
Procedure: ostap — this block is performed under general anesthesia in this patients for postoperative analgesia.
  Groups: OSTAP
Procedure: SIPB plus rectus sheath block — this block is performed under general anesthesia in this patients for postoperative analgesia.
  Groups: SIPB plus rectus sheath block

SUMMARY:
the investigators use usually a plane block for postoperative analgesia; if it suitable. İn laparoscopic patients; investigators used oblique subcostal transversus abdominis plane block; formerly. But in the last few months, the investigators have performed serratus intercostal (BRILMA) block with bilateral rectus sheath block. in this retrospective evaluation, the aim of the retrospective evaluation is to determine the effects of two block on postoperative opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoed laparoscopic cholecystectomy ASA I-II-III

Exclusion Criteria:

* patients used another block or block combination
* no block performed patients
* procedure converted to open procedure

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult patients undergoing laparoscopic cholecystectomy, ASA I-II-III patients.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-26 (Actual)

PRIMARY OUTCOMES:
opioid consumption | 24 hours
  Tramadol consumption in Patient Controlled Analgesia device and additional and rescue analgesic using

SECONDARY OUTCOMES:
Pain assessed by NRS | 24 hours
  Changes in Numeric Rating Scale (NRS) at rest and on movement will be recorded at intervals. NRS is a unidimensional measure of pain intensity in adults. The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

CONTACTS AND LOCATIONS:
Overall Officials: serkan tulgar, Principal Investigator — Maltepe University
Locations (1):
- Maltepe University faculty of medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen Y, Shi K, Xia Y, Zhang X, Papadimos TJ, Xu X, Wang Q. Sensory Assessment and Regression Rate of Bilateral Oblique Subcostal Transversus Abdominis Plane Block in Volunteers. Reg Anesth Pain Med. 2018 Feb;43(2):174-179. doi: 10.1097/AAP.0000000000000715. PMID 29278604
- [Background] Fernandez Martin MT, Lopez Alvarez S, Perez Herrero MA. Serratus-intercostal interfascial block as an opioid-saving strategy in supra-umbilical open surgery. Rev Esp Anestesiol Reanim (Engl Ed). 2018 Oct;65(8):456-460. doi: 10.1016/j.redar.2018.03.007. Epub 2018 May 20. English, Spanish. PMID 29789137